CLINICAL TRIAL: NCT05586243
Title: MAGNETIC RESONANCE SPECTROSCOPY BIOMARKERS IN TYPE 3 GAUCHER DISEASE (GD3)
Status: Recruiting | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: MEDICAL PROTOCOL (HRP-590)
Record Dates: First submitted 2022-10-16; First posted 2022-10-19 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Gaucher Disease, Type 3
MeSH Terms: conditions — Gaucher Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — During the visit, participants will undergo a blood sample collection. Blood sample will be processed and stored for future analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — This is an observational study looking at brain chemicals related to oxidative stress and inflammation using magnetic resonance spectroscopy (MRS).

SUMMARY:
Recent studies have has shown that magnetic resonance spectroscopy (MRS) can provide validated neuronal markers in patients with Type 1 GD (GD1) who are on stable therapy. However, alterations in neurometabolites in adult patients with GD3, who have established neurological involvement, are not well understood. The goal of this study is to characterize neurometabolite profiles in adult patients with GD3 using MRS to identify novel biomarkers that can demonstrate treatment response. Additionally, a secondary aim is to evaluate relationships between neurometabolites and disease parameters, such as genotype, enzyme levels and Gaucher disease (GD) biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* All participants must be 18 years or older.
* All enrollees must understand and cooperate with requirements of the study in the opinion of the investigators and must be able to provide written informed consent.
* Individuals with GD3 who are medically stable for participation in study in the opinion of the investigator.

Exclusion Criteria:

* Medically unstable conditions as determined by the investigators.
* Concurrent disease; medical condition; or an extenuating circumstance that, in the opinion of the investigator, might compromise subject safety, study compliance, completion of the study, or the integrity of the data collected for the study.
* Women who are pregnant or lactating or of child-bearing age that are not using acceptable forms of contraception.
* Patients enrolled in another interventional study.
* Patients who cannot or are unwilling to have blood drawn.
* Inability to undergo Magnetic Resonance Imaging (MRI) scanning, including but not limited to unable to remain still in an MRI scanner for more than 30 minutes, claustrophobia, presence of paramagnetic substances or pacemakers in body, weight over 300 lbs.
* Unable to adhere to study protocol for whatever reason.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants with GD3
Sampling Method: Non-Probability Sample
Enrollment: 5 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Neurometabolite profile | baseline
  Characterize neurometabolite profiles of up to 18 metabolites including N-acetyl aspartate (a validated biomarker of neuronal integrity), glutamate and GABA (neurotransmitters), myo-inositol, glutamine, lactate and choline (inflammation biomarkers) and glutathione (anti-oxidant) in individuals with GD3.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No